CLINICAL TRIAL: NCT07030322
Title: Health and Financial Impact on the Use of a Personal Exoskeleton in the Home and Community: a Case Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Ekso Bionics (Industry)
Responsible Party: Sponsor
Other Study IDs: 1385701
Record Dates: First submitted 2025-05-30; First posted 2025-06-22 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury
Keywords: exoskeleton; spinal cord injury; SCI; healthcare spending
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects with spinal cord Injury (SCI) who have a personal overground robotic exoskeleton device: Adults with a medical diagnosis of a spinal cord injury and sufficient upper extremity strength to manage approved stability aids (crutches, walker) who have access to a robotic exoskeleton device (Ekso Indego Personal) for use at home and in the community.
  Interventions: Device: Overground Robotic Exoskeleton

INTERVENTIONS:
Device: Overground Robotic Exoskeleton — Participants will have received training on their personal exoskeleton device prior to data collection. There is no required use dosage of the Ekso Indego Personal for this observational study.

SUMMARY:
The goal of this clinical trial is to examine the long-term use of a personal overground robotic exoskeleton in subjects with spinal cord injury. The main aims of this study include:

1. Determine patterns of personal overground robotic exoskeleton use over 12 months.
2. Examine the impact of personal overground robotic exoskeleton use on health outcomes over 12 months. These will include:

   1. Objective health - heart rate, physical activity, sleep behavior, body temperature, body-mass index, and bone density
   2. Medical status - rehospitalization, infection frequency, pressure injury, falls, fractures, medication (type/dose)
   3. Function - bowel function, bladder function, pain, spasticity, quality of life, mental health, social participation
3. Determine healthcare expenditure over 12 months

Participants and their support person(s) will be trained on using a personal robotic exoskeleton in their home and community. Once they complete training, they will use the exoskeleton as they wish (ie, no requirement to use the device a certain number of times per week) and data collection will begin.

DETAILED DESCRIPTION:
This prospective observational study will recruit and enroll individuals with SCI. These individuals will be part of a convenience sample due to employment or volunteer work with Ekso Bionics. They will be own or have access to an Indego Personal exoskeleton for home use. The parallel mixed methods design will allow for quantitative and qualitative data collected concurrently and integrated with equal consideration. Eligible individuals will be identified through work with representatives at Ekso Bionics for device acquisition and set up of training. Individuals who acquire a personal device will be screened for eligibility (criteria detailed below) and qualifying patients will be approached to participate. Upon providing consent, participants will complete quantitative and qualitative assessments over 12 months. Assessments will be conducted on five occasions: (1) baseline, (2) 1-month post-enrollment, (3) 3-months post-enrollment, (4) 6-months post-enrollment, and (5) 12-months post-enrollment. All study specific assessments will be completed by trained assessors. Quantitative and qualitative assessments will be completed by a physical therapist or other member of the research staff with necessary training. Time commitment for each participant at each assessment is 60 to 90 minutes.

Additionally, participants will be fitted for and provided at study enrollment with a wearable medical monitoring device for continuous tracking over 12-months. Study staff will provide each participant with a personal device account, to be set up using a premade study email, during enrollment. These emails will be generated utilizing a unique identifier feature which allows a single email to be suffixed with a unique identifier (e.g., study email account: "EksoIndegoStudy@gmail.com", participant S001 Wearable sensor account: "EksoIndegoStudy+S001@gmail.com"). Each account will be linked to a research data collection platform at Ekso Bionics. Ekso Bionics will collect necessary data from the wearable sensors including: heart rate, physical activity, sleep data, stress scores, weight, and profile information. To maintain blinding of potential health data, we will use the 1st of the birth month for each participant, so activity levels based on age can still be calculated appropriately. Data from the wearable device will be retrieved from the manufacturer cloud-based storage. All data is available for export by study staff either individually or as batch data, including all de-identified participant data in one file.

No specific intervention will take place during this observational study. However, each will have access to an Ekso Indego Personal device for home and community use. The Ekso Indego Personal (Indego) is a wearable powered exoskeleton device that actively assists individuals to stand and walk; these are individuals with walking impairments resulting from lower extremity weakness or paralysis due to spinal cord injury. Unique in design, the Indego consists of five (5) snap-together components (the lumbar/hip section, right and left upper leg sections, and right and left lower leg sections). The hip component houses a rechargeable battery pack, while each upper leg component houses two motors as well as embedded sensors and controllers. The Ekso Indego Personal incorporates powered movement of both hip and knee joints, in addition to built-in ankle-foot-orthoses (AFOs) at both ankle joints, which provide ankle support and stability, and also transfers the weight of the exoskeleton to the ground. The Ekso Indego Personal requires use of a stability aid, such as a rolling walker or set of forearm crutches. Once acquired, participants will complete device training and utilize their personal Ekso Indego exoskeleton according to their individual preferences with their certified support person.

Assessments will include: brief usage survey, 1-1 focused interview on device usage, device data, objective health data captured by wearable health monitor, self-reported BMI, bone mineral density, medical status questionnaire, Modified International SCI Lower Urinary Tract Function Basic Data Set, Modified International SCI Bowl Function Basic Data Set, pain questionnaire, Penn Spasm Frequency Scale, quality of life questionnaire, General Anxiety Disorder-7, Craig Handicap Assessment And Reporting Technique, health encounters survey, 1-1 focused interview on healthcare encounters, and medical records review.

ELIGIBILITY:
Inclusion Criteria:

* Femur lengths from 14.5" to 19" (35.5cm to 47 cm)
* Healthy bone density
* Height from 5'1" to 6'3" (1.5 to 1.9 m)
* Seated hip width ≤ 16.6" (42.2 cm)
* Sufficient upper extremity strength to manage approved stability aids
* Weight 250 lbs or less
* Availability of a support person able to complete training and be present during all Indego sessions

Exclusion Criteria:

* Cognitive impairments resulting in inability to follow directions
* Colostomy bag
* Diminished standing tolerance caused by orthostatic hypotension
* Heterotopic ossification
* Hip or knee contractures greater than 10° or ankle contractures greater than 5°
* History of severe neurological injuries other than SCI (multiple sclerosis, --cerebral palsy, amyotrophic lateral sclerosis, traumatic brain injury, etc).
* Lower limb prothesis
* Poor skin integrity in areas in contact with the device
* Pregnancy
* Psychiatric conditions that may interfere with proper operation of the device
* Severe concurrent medical diseases: infections, circulatory, heart or lung, pressure sores
* Severe or uncontrolled spasticity (Modified Ashworth 4)
* Spinal instability or spinal orthotics
* Uncontrolled autonomic dysreflexia
* Uncontrolled hypertension or hypotension
* Unhealed limb or pelvic fractures
* Unresolved deep vein thrombosis
* Any condition which in the opinion of a medical doctor prevents the user from using the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ekso Bionics Clinical team will identify ambassadors with SCI who are interested in attaining an Indego device.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in sessions recorded and provided by the exoskeleton device across study timepoints | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Indego device records and transmits electronically data regarding each session completed on device. These include the number of sessions, total number of steps, total time spent with device on, and total time spent walking. For each individual Indego session: number of steps, time of session, and time spent walking. From the last study checkpoint, the shortest time spent walking and longest time spent walking will also be recorded.
  Use habits will be recorded over the duration of the study from baseline to 12-months post-enrollment and it will be determined if use increases over time, decreases over time, or remains consistent. This outcome will address total and average number of Indego sessions completed per month.
Change in time spent walking recorded and provided by the exoskeleton device across study timepoints | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Indego device records and transmits electronically data regarding each session completed on device. These include the number of sessions, total number of steps, total time spent with device on, and total time spent walking. For each individual Indego session: number of steps, time of session, and time spent walking. From the last study checkpoint, the shortest time spent walking and longest time spent walking will also be recorded.
  Use habits will be recorded over the duration of the study from baseline to 12-months post-enrollment and it will be determined if use increases over time, decreases over time, or remains consistent. This outcome measures average time spent walking per month measured in hours:minutes:seconds.
Change in walking time recorded and provided by the exoskeleton device across study timepoints | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Indego device records and transmits electronically data regarding each session completed on device. These include the number of sessions, total number of steps, total time spent with device on, and total time spent walking. For each individual Indego session: number of steps, time of session, and time spent walking. From the last study checkpoint, the shortest time spent walking and longest time spent walking will also be recorded.
  Use habits will be recorded over the duration of the study from baseline to 12-months post-enrollment and it will be determined if use increases over time, decreases over time, or remains consistent. This outcome will measure total and average walking time in the Indego per month measured in hours:minutes:seconds.
Change in usage metrics as reported by user | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Indego device records and transmits electronically data regarding each session completed on device. These include the number of sessions, total number of steps, total time spent with device on, and total time spent walking. For each individual Indego session: number of steps, time of session, and time spent walking. From the last study checkpoint, the shortest time spent walking and longest time spent walking will also be recorded.
  Use habits will be recorded over the duration of the study from baseline to 12-months post-enrollment and it will be determined if use increases over time, decreases over time, or remains consistent. This outcome will ask participant(s) if they feel like they are using their device more/less/same as last timepoint.
Change in medical health status, assessed by interview and written questions based on the SCI Model Systems form II, between all timepoints in study | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Utilized the SCI Model Systems form II as a guide, questions will be asked to assess medical health status at each timepoint. These questions ask the participant(s) to rate their current health from poor to excellent and any changes in health since last checkpoint on a scale from much worse now to much better now. Number of falls, fractures, urinary tract infections, hospitalizations, healthcare visits, and emergency room visits will also be collected. For hospitalizations, healthcare visits, and emergency room visits, purpose of each will be collected. Medications will be collected including name, frequency, and dose. This information will be gathered at each checkpoint and compared for changes between timepoints but also between baseline and 12-month post enrollment.
Change in bladder function between 5 timepoints using the Modified International SCI Lower Urinary Tract Function Basic Data set | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Modified International SCI Lower Urinary Tract Function Basic Data set is created by the International Spinal Cord Society to standardize the collection information on the lower urinary tract in daily clinical practice. This is not a scored outcome, and is instead a set of standardized questions. Questions examine how the bladder is emptied, average number of emptying, incontinence, medication usage, and surgical procedures related to bladder. Any changes in these answers over the course of the 12-month study will be recorded and analyzed.
Change in bowel function between 5 timepoints using the Modified International SCI Bowel Function Basic Data set | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Modified International SCI Bowel Function Basic Data set is created by the International Spinal Cord Society to standardize the collection information on bowel function in daily practice. This is not a scored outcome, and is instead a set of standardized questions. Data collected includes any surgical procedures on the gastrointestinal tract, defecation method, average time to defecate, frequency of defecation, incontinence, tools/medications utilized to help manage bowel, and abdominal pain. Any changes in these answers over the course of the 12-month study will be recorded and analyzed.
Changes in pain between 5 timepoints in study measured by questions from SCI Model Systems Form II | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Pain intensity on a scale of 0-10 with 0 meaning no pain and 10 meaning severe pain, location of pain, description of pain (including options of shooting, constant, burning, tingling, among others) and pain's interference in normal work rated from not at all to extreme interference will be examined . These questions are based off questions from the SCI Model Systems form II which standardizes how we collect data on this topic. Any changes between baseline and any time point (1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment) will be recorded and analyzed
Changes in spasticity from baseline to 4 other timepoints in study measured by Penn Spasm Frequency Scale | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Penn Spasm Frequency Scale is a self-report measure used to assess a patient's perception of spasticity frequency and severity. This scale has excellent internal consistency. Participants will be asked to rate their frequency of spasms on a scale of 0 (no spasms) to 4 (occurring more than 10 times per hour) and the spasm severity on a scale of 1 (mild) to 3 (severe). Any changes between baseline and any time point (1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment) will be recorded and analyzed.
Change in quality of life assessed by the SCI Model Systems form II SCI-QOL and Satisfaction with Life scale from baseline to 4 other time points during study | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Quality of life will be assessed by questions from the SCI Model Systems Form II SCI-QOL Resilience short form, which asks 8 questions each rated from never to always. The satisfaction with life scale, also from which the SCI model Systems Form II, asks 5 questions where the participant(s) rates how much they agree or disagree with each statement. Total scores will be calculated for each scale, where in both scales, lower total scores correlate to lower QOL. Any changes between baseline and other measurement time points will be collected and analyzed.
Change in mental health measured by general anxiety disorder (GAD-7) between baseline and 4 other data collection points over 12 months | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  The GAD-7 is recommended by National Institute of Neurologic Disorders and Stroke Spinal Cord Injury Common Data Elements (NINDS SCI CDE) and used by the spinal cord injury (SCI) Model Systems, the GAD-7 assesses the anxiety of our participants with SCI. Consists of seven questions assessing how often the subject has been bothered by these items over the last 2 weeks, each scaled from 0 (not at all sure) to 3 (nearly every day). A total score of 5 is classified as mild anxiety, 10 is classified as moderate anxiety, and 15 is classified as severe anxiety. This measure has high sensitivity and specificity. It will be taken at baseline and 4 other study timepoints and changes between each assessment will be analyzed.
Change in participation between baseline and 4 other study timepoints measured by the Craig Handicap Assessment And Reporting Technique (CHART) | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  The Craig Handicap Assessment And Reporting Technique (CHART) is administered through long form document. Subscales for physical independence, cognitive independence, mobility, occupation, social integration, and economic self sufficiency are scored independently. Each subscale is scored out of 100, which indicates no handicap in that section. Lower scores indicate greater handicap in that section. Any changes in subscale scores between baseline and 4 other time points will be analyzed.
Compare healthcare expenditure from 12 months prior to exoskeleton initiation (baseline) and the year following exoskeleton acquisition by examining medical and billing records | retrospective analysis of 12 months prior to exoskeleton acquisition, 12 months following completion of training on exoskeleton device
  Medical and Billing records for a total of 24 months (12 months prior to exoskeleton acquisition and the 12 months following completion of exoskeleton training) will be collected for each subject. Total healthcare expenditure costs will be compared between the two 12-month periods. Cost of each healthcare visit, emergency room visit, and hospital admission will be calculated. Medication cost per refill and supply costs (example: catheters) will be calculated and compared year over year. Costs will also be broken down into subcategories including hospitalizations, wound-related, bowel/bladder related, medication, etc.
Change in participant satisfaction regarding use of exoskeleton | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Both written and interview questions will be posed to the participant to assess their impression regarding their Indego usage. Questions will assess if participant has had any issues with their Indego, are they happy with the number sessions they are using their Indego and the length of each session, what activities the participant is using the Indego for, the biggest reason for not using the Indego more often and for longer, and how the participant perceives their use compared to the last checkpoint. These answers will be qualitative and recorded at five checkpoints during the study.
Frequency of adverse events (AEs) and serious adverse events (SAEs) throughout 12 month study | Through study completion, 1 year
  AEs and SAEs will be tracked throughout the 12 months of the study. An adverse event form will be filled out for each AE or SAE which will include a description of the event, the action taken (medications, procedure, etc), duration of the event, if it was related to the Indego and/or the study protocol, and classification of the event. Number of events will be calculated throughout the study and reported on.

SECONDARY OUTCOMES:
Changes in heart rate measured by wearable health monitoring device from baseline to study completion | Through study completion, 1 year
  A wearable health monitoring device (Oura ring) will be provided to each study participant. Each participant will be asked to wear this device at all times throughout the 12-month study duration except when it is charging. The following heart rate data will be collected: daytime lowest average heartrate (HR) per day, daily time in restorative HR, daily time in stress HR zone, sleep HR range high, sleep HR range low, resting heart rate, and heart rate variability. Data will be graphed over the full year of the study (baseline to 12 months post) and trends assessed, with specific interest on change from baseline to 12-month post.
Change in sleep behavior over the duration of the 12-months using a wearable health monitoring device | Through study completion, 1 year
  Each participant will be fitted with a wearable health monitoring system (Oura ring) that they will be instructed to wear at all times when it is not charging. This device will track sleep, including time awake per day, time in REM per day, time in light sleep per day, time in deep sleep per day, average sleep time per week, and sleep score per day. This information will be graphed throughout the 12 month study period and trends will be tracked. Change in each value between baseline and 12-month post enrollment will be calculated.
Change in body temperature over the duration of the 12-months using a wearable health monitoring device | Through study completion, 1 year
  Each participant will be fitted with a wearable health monitoring system (Oura ring) that they will be instructed to wear at all times when it is not charging. This device will track body temperature average per day. The amount above or below temperature baseline will be collected per day. Data will be collected and graphed over the entire duration of the 12-month study. Trends in body temperature fluctuation will be assessed. Change from baseline to 12-month post enrollment will be calculated.
Changes in body mass index (BMI) at 5 time points during the study based on self reported height and weight | baseline, 1-month post-enrollment, 3-months post-enrollment, 6-months post-enrollment, and 12-months post-enrollment.
  Subjects will be asked to self-report height and weight at 5 time points during the 12-month study. BMI will be calculated by dividing weight in kilograms by height in meters squared. BMI values of less than 18.5 are categorized as underweight, those with BMI from 18.5 to 24.9 are categorized as being healthy weight, those with BMI from 25 to 29.9 are categorized as overweight, and those with BMI of 30 or more are categorized as obese. Changes in BMI will be analyzed as well as any change in BMI category.
Change in bone mineral density (BMD) will be assessed using dual-energy x-ray absorptiometry (DXA) at baseline and conclusion of the study with comparison of z scores assessed. | baseline and 12-months post-enrollment
  DXA scan will be completed at baseline and conclusion of the study and z scores compared. DXA scans are a common part of spinal cord injury healthcare to help determine if the long bones in the legs are able to sustain the weight of the body in a standing position. While there are no formal cut-off scores, recommended guidelines for BMD for safe walking with the exoskeleton are a Z score less than -2. Change in z score from baseline to 12-month post enrollment will be calculated.
Changes in heart rate during exercise sessions using Indego from baseline to 12-month post enrollment | Through study completion, 1 year
  A wearable health monitoring device (Oura ring) will be provided to each study participant. Each participant will be asked to wear this device at all times throughout the 12-month study duration except when it is charging. Heart Rate data will be extrapolated for each time period when participant is in the exoskeleton with focus on highest and lowest heartrate values during the period of walking in the Indego. Highest and lowest exercise heartrate will be graphed over the full 12 months and a comparison from baseline to 12-month post enrollment will be calculated.
Change in number of steps per day over the duration of the 12-months using a wearable health monitoring device | Through study completion, 1 year
  Each participant will be fitted with a wearable health monitoring system (Oura ring) that they will be instructed to wear at all times when it is not charging. This device will record daily steps. Data will be collected and graphed over the entire duration of the 12-month study. Trends in steps per day will be assessed. Change from baseline to 12-month post enrollment will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ekso Bionics, Inc., San Rafael, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorman PH, Forrest GF, Asselin PK, Scott W, Kornfeld S, Hong E, Spungen AM. The Effect of Exoskeletal-Assisted Walking on Spinal Cord Injury Bowel Function: Results from a Randomized Trial and Comparison to Other Physical Interventions. J Clin Med. 2021 Mar 2;10(5):964. doi: 10.3390/jcm10050964. PMID 33801165
- [Background] Baunsgaard CB, Nissen UV, Brust AK, Frotzler A, Ribeill C, Kalke YB, Leon N, Gomez B, Samuelsson K, Antepohl W, Holmstrom U, Marklund N, Glott T, Opheim A, Penalva JB, Murillo N, Nachtegaal J, Faber W, Biering-Sorensen F. Exoskeleton gait training after spinal cord injury: An exploratory study on secondary health conditions. J Rehabil Med. 2018 Sep 28;50(9):806-813. doi: 10.2340/16501977-2372. PMID 30183055
- [Background] Priebe MM, Sherwood AM, Thornby JI, Kharas NF, Markowski J. Clinical assessment of spasticity in spinal cord injury: a multidimensional problem. Arch Phys Med Rehabil. 1996 Jul;77(7):713-6. doi: 10.1016/s0003-9993(96)90014-3. PMID 8670001
- [Background] Hsieh JT, Wolfe DL, Miller WC, Curt A; SCIRE Research Team. Spasticity outcome measures in spinal cord injury: psychometric properties and clinical utility. Spinal Cord. 2008 Feb;46(2):86-95. doi: 10.1038/sj.sc.3102125. Epub 2007 Oct 2. PMID 17909559
- [Background] Krogh K, Emmanuel A, Perrouin-Verbe B, Korsten MA, Mulcahey MJ, Biering-Sorensen F. International spinal cord injury bowel function basic data set (Version 2.0). Spinal Cord. 2017 Jul;55(7):692-698. doi: 10.1038/sc.2016.189. Epub 2017 Feb 14. PMID 28195229
- [Background] Biering-Sorensen F, Kennelly M, Kessler TM, Linsenmeyer T, Pannek J, Vogel L, Wyndaele JJ. International Spinal Cord Injury Lower Urinary Tract Function Basic Data Set (version 2.0). Spinal Cord Ser Cases. 2018 Jul 6;4:60. doi: 10.1038/s41394-018-0090-7. eCollection 2018. PMID 30002915
- [Background] Shackleton C, Evans R, West S, Derman W, Albertus Y. Robotic Walking to Mitigate Bone Mineral Density Decline and Adverse Body Composition in Individuals With Incomplete Spinal Cord Injury: A Pilot Randomized Clinical Trial. Am J Phys Med Rehabil. 2022 Oct 1;101(10):931-936. doi: 10.1097/PHM.0000000000001937. Epub 2021 Dec 6. PMID 34864766
- [Background] Abdelrahman S, Ireland A, Winter EM, Purcell M, Coupaud S. Osteoporosis after spinal cord injury: aetiology, effects and therapeutic approaches. J Musculoskelet Neuronal Interact. 2021 Mar 1;21(1):26-50. PMID 33657753
- [Background] Cahill A, Ginley OM, Bertrand C, Lennon O. Gym-based exoskeleton walking: A preliminary exploration of non-ambulatory end-user perspectives. Disabil Health J. 2018 Jul;11(3):478-485. doi: 10.1016/j.dhjo.2018.01.004. Epub 2018 Feb 1. PMID 29500092
- [Background] van Dijsseldonk RB, van Nes IJW, Geurts ACH, Keijsers NLW. Exoskeleton home and community use in people with complete spinal cord injury. Sci Rep. 2020 Sep 24;10(1):15600. doi: 10.1038/s41598-020-72397-6. PMID 32973244
- [Background] Sikka S, Callender L, Driver S, Bennett M, Reynolds M, Hamilton R, Warren AM, Petrey L. Healthcare utilization following spinal cord injury: Objective findings from a regional hospital registry. J Spinal Cord Med. 2019 Mar;42(2):194-200. doi: 10.1080/10790268.2018.1505330. Epub 2018 Oct 2. PMID 30277845
- [Background] Skelton F, Hoffman JM, Reyes M, Burns SP. Examining health-care utilization in the first year following spinal cord injury. J Spinal Cord Med. 2015 Nov;38(6):690-5. doi: 10.1179/2045772314Y.0000000269. Epub 2014 Oct 9. PMID 25299152
- [Background] Stillman MD, Frost KL, Smalley C, Bertocci G, Williams S. Health care utilization and barriers experienced by individuals with spinal cord injury. Arch Phys Med Rehabil. 2014 Jun;95(6):1114-26. doi: 10.1016/j.apmr.2014.02.005. Epub 2014 Feb 22. PMID 24565745
- [Background] Cardenas DD, Hoffman JM, Kirshblum S, McKinley W. Etiology and incidence of rehospitalization after traumatic spinal cord injury: a multicenter analysis. Arch Phys Med Rehabil. 2004 Nov;85(11):1757-63. doi: 10.1016/j.apmr.2004.03.016. PMID 15520970
- [Background] Fogelberg D, Atkins M, Blanche EI, Carlson M, Clark F. Decisions and Dilemmas in Everyday Life: Daily Use of Wheelchairs by Individuals with Spinal Cord Injury and the Impact on Pressure Ulcer Risk. Top Spinal Cord Inj Rehabil. 2009 Fall;15(2):16-32. doi: 10.1310/sci1502-16. PMID 21603085
- [Background] Jensen MP, Truitt AR, Schomer KG, Yorkston KM, Baylor C, Molton IR. Frequency and age effects of secondary health conditions in individuals with spinal cord injury: a scoping review. Spinal Cord. 2013 Dec;51(12):882-92. doi: 10.1038/sc.2013.112. Epub 2013 Oct 15. PMID 24126851
- [Background] Louie DR, Eng JJ, Lam T; Spinal Cord Injury Research Evidence (SCIRE) Research Team. Gait speed using powered robotic exoskeletons after spinal cord injury: a systematic review and correlational study. J Neuroeng Rehabil. 2015 Oct 14;12:82. doi: 10.1186/s12984-015-0074-9. PMID 26463355
- [Background] Tefertiller C, Hays K, Jones J, Jayaraman A, Hartigan C, Bushnik T, Forrest GF. Initial Outcomes from a Multicenter Study Utilizing the Indego Powered Exoskeleton in Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2018 Winter;24(1):78-85. doi: 10.1310/sci17-00014. Epub 2017 Nov 20. PMID 29434463
- [Background] Sale P, Franceschini M, Waldner A, Hesse S. Use of the robot assisted gait therapy in rehabilitation of patients with stroke and spinal cord injury. Eur J Phys Rehabil Med. 2012 Mar;48(1):111-21. PMID 22543557
- [Background] Chen G, Chan CK, Guo Z, Yu H. A review of lower extremity assistive robotic exoskeletons in rehabilitation therapy. Crit Rev Biomed Eng. 2013;41(4-5):343-63. doi: 10.1615/critrevbiomedeng.2014010453. PMID 24941413
- [Background] Esquenazi A, Talaty M, Jayaraman A. Powered Exoskeletons for Walking Assistance in Persons with Central Nervous System Injuries: A Narrative Review. PM R. 2017 Jan;9(1):46-62. doi: 10.1016/j.pmrj.2016.07.534. Epub 2016 Aug 24. PMID 27565639
- [Background] Mekki M, Delgado AD, Fry A, Putrino D, Huang V. Robotic Rehabilitation and Spinal Cord Injury: a Narrative Review. Neurotherapeutics. 2018 Jul;15(3):604-617. doi: 10.1007/s13311-018-0642-3. PMID 29987763
- [Background] Mehrholz J, Pohl M. Electromechanical-assisted gait training after stroke: a systematic review comparing end-effector and exoskeleton devices. J Rehabil Med. 2012 Mar;44(3):193-9. doi: 10.2340/16501977-0943. PMID 22378603